CLINICAL TRIAL: NCT03463941
Title: Peer Support Dyads in a Health Promotion Program in African American Churches
Brief Title: Peer Support Dyads in Churches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00091547; 1F31NR017813-01 (NIH)
Record Dates: First submitted 2018-03-07; First posted 2018-03-13 (Actual); Results first posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Peer Support and Chronic Disease; Obesity; Type II Diabetes; Cardiovascular Disease; Cancer
Keywords: African American; Faith institutions; Dyads; Health disparities
MeSH Terms: conditions — Chronic Disease; Obesity; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- African American church members (Experimental)
  Interventions: Behavioral: Peer Support Dyad Intervention

INTERVENTIONS:
Behavioral: Peer Support Dyad Intervention — Phase I: At baseline and at post-intervention, participant height, weight, BMI, fruit and vegetable intake and exercise habits will be measured. Participants will complete surveys and meet each week to learn about nutrition and exercise.
  Phase II: Dyads will attend a communication training session to discuss 1) benefits of working with a partner; 2) supportive communication tips; and 3) expected activities for the next 8 weeks, including filling out daily logs. After the training session, the dyads will work together to achieve their health goals. The dyads will return to the church for two check in sessions. At these sessions, participants will turn in their logs, and be weighed. At the end of the intervention, BMI will be reassessed, and surveys and interviews will be completed.

SUMMARY:
The purpose of this study is to explore how working with a partner can influence participation in a church wellness program. There are many different types of church wellness programs. Church members are more likely to participate and achieve goals in these programs when they have peer support. The researcher would like to know what African American men and women think about working with a support partner. This information will help researchers design better church wellness programs. The participants are being asked to take part in this research because the investigators believe that it is helpful to share feelings and thoughts about experiences working with a partner to achieve health goals. This knowledge will be used to create church wellness programs that will help African American men and women prevent disease and live healthier lives.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria will be churches with mostly African American members.
* Participant criteria will be: ages >=18 or older who identify as African American
* Attend church at least once per week
* Speak, read and write English
* Willing to complete study activities and assessments
* Able to engage in moderate physical activity. (e.g., walking - based on their own activity level and assessment).

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Lipkus, Principal Investigator — Duke University
Locations (1):
- Faithful Families Program, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | African American Church Members
Started | 80
Completed | 62
Not Completed | 18

BASELINE CHARACTERISTICS:
Arm/Group | African American Church Members
Number analyzed (Participants) | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 44
  >=65 years | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 80
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 80
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.9 (7.2)
Weight [Mean (Standard Deviation); unit: pounds] | 198 (51.2)
Fruit and Vegetable Intake [Count of Participants; unit: Participants] — Number of participants consuming 7 or more fruits and vegetables per day.
  Participants | 1
Days of Physical Activity [Mean (Standard Deviation); unit: days] | 3.1 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Measured by Retention
Description: Retention will be calculated from the number of participants who continue to Phase II out of the number who complete Phase I (>50% attendance), and the attrition rate.
Time Frame: Baseline to week 18
Population: Participants who completed Phase I (>50% attendance).
Measure: Count of Participants; unit: Participants
Arm/Group | African American Church Members
Number analyzed (Participants) | 65
Participants | 62
Statistical Analysis 1: Comparison: African American Church Members; Test type: Other; descriptive

2. Primary Outcome: Number of Participants Who Agreed That Program Component Was Acceptable
Description: Measured by ten item feasibility survey, scored based on 5-point Likert scale administered at week 18, the last week of the program. Feasibility was measured on a scale of 1-5, where 1=strongly disagree that program component was acceptable or feasible, and 5=strongly agree that program component was acceptable or feasible)
Time Frame: Measured at Week 18
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | African American Church Members
Number analyzed (Participants) | 62
Participants | 61
Statistical Analysis 1: Comparison: African American Church Members; Test type: Other; descriptive

3. Primary Outcome: Health Educators' Perceptions of Feasibility as Measured by Semi-structured Interviews
Description: Reported as number of health educators who found the program to be feasible.
Time Frame: Measured at Week 18
Population: Health educators who were interviewed.
Measure: Count of Participants; unit: Participants
Groups:
- Health Educators: North Carolina Cooperative Extension nutrition educators who deliver the Faithful Families Thriving Communities curriculum to the faith community.
Arm/Group | Health Educators
Number analyzed (Participants) | 4
Participants | 4

4. Secondary Outcome: Goal Attainment as Measured by BMI (Body Mass Index)
Description: Mixed models will be used to assess changes in participant BMI pre and post intervention.
Time Frame: Week 18
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | African American Church Members
Number analyzed (Participants) | 62
kg/m^2 | 32 (6.8)
Statistical Analysis 1: Comparison: African American Church Members; Test type: Other; p < 0.05, Mixed Models Analysis

5. Secondary Outcome: Goal Attainment as Measured by Weight in Pounds
Description: A mixed model using intraclass correlation will be used used to assess changes in participant weight pre and post intervention.
Time Frame: Week 18
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | African American Church Members
Number analyzed (Participants) | 62
pounds | 189 (44.5)
Statistical Analysis 1: Comparison: African American Church Members; Test type: Other; p < 0.05, Mixed Models Analysis

6. Secondary Outcome: Goal Attainment as Measured by Number of Participants Consuming 7 or More Fruits and Vegetables Per Day
Description: A mixed model using intraclass correlation will be used to assess changes in participant fruit and vegetable intake pre and post intervention.
Time Frame: Week 18
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | African American Church Members
Number analyzed (Participants) | 62
Participants | 6
Statistical Analysis 1: Comparison: African American Church Members; Test type: Other; descriptive

7. Secondary Outcome: Goal Attainment as Measured by Days Per Week That Participants Exercised for 30 Minutes or More
Description: A mixed model using intraclass correlation will be used to assess changes in physical activity at weeks 1 and 18 pre and post intervention.
Time Frame: Week 18
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | African American Church Members
Number analyzed (Participants) | 62
days | 4.5 (2.2)
Statistical Analysis 1: Comparison: African American Church Members; Test type: Other; p < 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Baseline to 18 weeks
Arm/Group | African American Church Members
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT03463941/Prot_SAP_000.pdf